CLINICAL TRIAL: NCT02379650
Title: RCT Assessing Hydroxychloroquine for Unexplained Recurrent Pregnancy Loss
Brief Title: Hydroxychloroquine (HCQ) for Recurrent Pregnancy Loss
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Testing required by FDA for IND approval was too expensive to move forward with conduct of the study.
Sponsor: University of Utah (Other)
Collaborators: Intermountain Health Care, Inc. (Other)
Responsible Party: Principal Investigator, Robert Silver, M.D., University of Utah
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 78134
Record Dates: First submitted 2015-02-28; First posted 2015-03-05 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Recurrent Pregnancy Loss; Miscarriage
MeSH Terms: conditions — Abortion, Spontaneous | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydroxychloroquine (HCQ) (Experimental): Subjects in the experimental arm will take 400 mg hydroxychloroquine pills every day, starting before they get pregnant and continuing until 36 weeks of pregnancy or until the pregnancy is over.
  Interventions: Drug: Hydroxychloroquine (HCQ)
- Placebo (Placebo Comparator): Subjects in the experimental arm will take placebo pills every day, starting before they get pregnant and continuing until 36 weeks of pregnancy or until the pregnancy is over.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine (HCQ)
  Other Names: Plaquenil®
  Arms: Hydroxychloroquine (HCQ)
Drug: Placebo
  Arms: Placebo

SUMMARY:
Recurrent pregnancy loss (RPL) affects 5% of couples trying to achieve parenthood. Most cases of RPL are unexplained and have no effective treatment to improve the likelihood of a pregnancy resulting in a live birth. This leads to significant patient and provider frustration and emotional stress. Hydroxychloroquine (HCQ) is a medication commonly used in pregnancy to treat autoimmune and connective tissue diseases such as systemic lupus erythematosus (SLE). This use has shown that HCQ is very safe in pregnancy. HCQ has anti-inflammatory and anti-thrombotic effects and thus may improve pregnancy outcomes in couples with unexplained RPL. Although some providers are already prescribing HCQ for unexplained RPL, a randomized controlled trial is necessary to determine the true efficacy and safety of this treatment. This study has the potential to establish support for a new treatment option for unexplained RPL.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 18 and older
* Planning conception and have experienced 2 or more unexplained pregnancy losses prior to 20 weeks gestation and no more than one live birth

Exclusion Criteria:

* Documented antiphospholipd antibodies
* Uterine malformation or parental chromosomal abnormality
* Known lupus or other medical conditions that require treatment with hydroxychloroquine outside of this study protocol
* Any medical contraindications to hydroxychloroquine or aspirin therapy, including liver or kidney disease, pregestational diabetes or known retinopathy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2019-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Live Birth | Duration of gestation (up to 42 weeks)
  Frequency of pregnancies resulting in live birth

SECONDARY OUTCOMES:
Adverse Pregnancy Outcomes | Duration of gestation (up to 42 weeks)
  Preterm birth, fetal growth restriction, stillbirth, placental insufficiency

CONTACTS AND LOCATIONS:
Overall Officials: Robert Silver, MD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - Intermountain Healthcare, Salt Lake City, Utah
  - University of Utah Hospital, Salt Lake City, Utah